CLINICAL TRIAL: NCT03383159
Title: Gut Microbiota Prediction of Metachronous Colorectal Neoplasms in Patients With Colorectal Cancer
Brief Title: Gut Microbiota Prediction of Metachronous Colorectal Neoplasms
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Yunwei Wei 2017-3
Record Dates: First submitted 2017-12-17; First posted 2017-12-26 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2017-10

CONDITIONS: Gut Microbiota; Metachronous Adenoma
Keywords: Microbiota; Metachronous Adenoma; Colorectal Cancer; Colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Human fecal samples for DNA extraction
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Observation group 1: Patients who suffered metachronous adenoma after proximal colorectum cancer surgery.
- Control group 1: Patients who do not suffere metachronous adenoma after proximal colorectum cancer surgery.
- Observation group 2: Patients who suffered metachronous adenoma after distal colorectum cancer surgery.
- Control group 2: Patients who do not suffered metachronous adenoma after distal colorectum cancer surgery.

SUMMARY:
Patients with colorectal cancer are known to be at high risk of developing metachronous adenoma, however, participation in colonoscopy are low. Colonoscopy, the primary modality used all over the word, is costly and invasive, and its efficacy depends on the endoscopist's skill and the patient's bowel preparation. As life expectancy of patients with history of colon cancer is increasing, colonoscopy would increase the overall cost for patients and for the health care system. This study aim to construct a predictive model of postoperative colorectal neoplasm development using microbiota analysis.

DETAILED DESCRIPTION:
Colorectal cancer(CRC) is one of the most common malignancies in China and in Western countries. Furthermore, those with a history of CRC are at a higher risk for developing metachronous adenomas or CRC recurrence during the followup period. It has been reported that 0.7% of patients develop metachronous CRC during the 3 years after surgical resection for the initial CRC.

Surveillance colonoscopy is highly recommended by major international scientific societies with the intent of either detecting anastomotic recurrence at an early, curable stage or identifying metachronous premalignant(ie, adenomas) and malignant lesions. As life expectancy of patients with history of colon cancer is increasing, the costly and invasive postoperative examination increased the overall cost and suffering for patients.

The human colon plays host to a diverse and metabolically complex community of microorganisms. While colonic microbiome development along the colorectal adenoma-carcinoma sequence. Investigators speculate that gut microbiota related to metachronous adenoma or CRC, after curative treatment.

This study aim to discover if any difference of gut microbiota exist in patients who suffer from metachronous adenomas compared with patients who do not. Further try to seek the divergence microbiota of metachronous adenomas between Proximal and Distal Colorectum. construct a predictive model of postoperative colorectal neoplasm development using microbiota analysis. Finally, using microbita construct a predictive model of postoperative colorectal neoplasm development.

ELIGIBILITY:
Inclusion Criteria:

* Requirements of informed consent and assent of participant, parent or legal guardian as applicable
* Patients who underwent exhaustive colorectal cancer surgical resection and accept colonoscopy
* Patients between the age of 35 and 75 years old without considering sex
* Patients with BMI= 18.5-23.9
* Participants can follow the visit plan

Exclusion Criteria:

* Patients with colorectal cancer with distant metastasis
* Chronic renal diseases and hepatic cirrhosis
* Chronic ischemic heart disease with unstable angina, chronic heart failure at class III or IV and acute myocardial infarction in the last 6 months
* Individuals with a history of Chronic diarrhea
* Individuals with a history of Diabetes mellitus
* Individuals with a history of Hypertension
* Individuals with a history of autoimmune diseases
* Use of antibiotics and probiotics 3 mouth before samples collection
* Individuals with a history of abdominal operation due to any reason
* Individuals with any history of cancer other than colorectal cancer
* Individuals with Inflammatory bowel disease

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients underwent an exhaustive colorectal cancer surgical resection in the First Affiliated Hospital of Harbin Medical University from December 1, 2012 to April 28, 2017. Each participant provided a fresh stool sample in hospital before bowel preparation or 1 month after colonoscopy. All patients did not use antibiotics and probiotics 3 mouth before samples collection.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-05-01 (Actual); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Differences In Microbiota | 1, 3 and 5 years after surgery
  The diversity, structure of microbiota and relative abundance of special bacterial taxa 16S rRNA gene sequencing will be performed.

SECONDARY OUTCOMES:
Predictive model establish | June to August of 2018
  Using microbita construct a predictive model of postoperative colorectal neoplasm development.
Predictive model validation | August of 2018 to April of 2019
  Validation the accuracy of the predictive model.

CONTACTS AND LOCATIONS:
Overall Officials: Yunwei Wei, Principal Investigator — First Affiliated Hospital of Harbin Medical University
Locations (1):
- First affiliated hospital of Harbin medical university, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No